CLINICAL TRIAL: NCT00323752
Title: Recombinant Human Erythropoietin Compared to Autologous Pre-Donation Prior to Scoliosis Surgery in Children.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Eleanor Reimer, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C02-0510; W02-0166
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Scoliosis
Keywords: Blood loss, Erythropoetin
MeSH Terms: conditions — Scoliosis; Hemorrhage

INTERVENTIONS:
Procedure: rHuEpo — Subjects will be randomly assigned to either participate in the PAD program or receive the rHuEpo treatment. Subjects in the PAD group will donate 1 unit of blood at -14 and -7 days prior to surgery. A dose of 500 IU of rHuEpo will be administered subcutaneously to subjects in the rHuEpo group at -21, -14, and -7 days prior to surgery.

SUMMARY:
The purpose of this study is to establish whether rHuEpo is as effective as PAD in increasing red cell mass prior to surgery. Other benefits of the PAD program and preoperative administration of rHuEpo will also be compared.

DETAILED DESCRIPTION:
Background The pre-operative autologous donation (PAD) program was established at British Columbia's Children's Hospital in 1988 to decrease the need for homologous blood transfusion. It could alleviate the constraints arising from current and expected future shortages of homologous blood. But, primarily, the introduction of PAD was driven by concern about blood borne diseases.

A patient's own blood is generally considered to be the safest blood. However, the PAD program has several shortcomings. Firstly, venous access for blood withdrawal is often difficult in children. Secondly, the PAD program at British Columbia's Children's Hospital (BCCH) has a history of considerable wastage. Approximately 50% of pre-donated blood is discarded. Thirdly, a patient's medical condition or distance from BCCH can make participation in the program infeasible. Finally, even though the donor and recipient are the same, PAD is still susceptible to bacterial contamination and clerical errors. For example, it is possible that the wrong blood, either homologous blood or another patient's autologous blood, may be given to the PAD donor or another patient.

Wastage, cost, logistic challenges, and safety concerns have driven our interest in an alternative treatment for scoliosis patients. Recombinant human erythropoietin (rHuEpo) is a hormone that stimulates red cell production. This treatment has been used for patients scheduled for scoliosis surgery since 1990. However, it is not part of BCCH's current practice.

Study Objectives The purpose of this study is to establish whether rHuEpo is as effective as PAD in increasing red cell mass prior to surgery. Other benefits of the PAD program and preoperative administration of rHuEpo will also be compared.

A pilot study of 20 subjects to investigate whether the gain in the PAD group is different from the group treated with rHuEpo..

Research Activities Females aged 12 to 18 years that are scheduled to undergo correction of idiopathic scoliosis by posterior fusion will be enrolled in the study. Subjects will be randomly assigned to either participate in the PAD program or receive the rHuEpo treatment. Subjects in the PAD group will donate 1 unit of blood at -14 and -7 days prior to surgery. A dose of 500 IU of rHuEpo will be administered subcutaneously to subjects in the rHuEpo group at -21, -14, and -7 days prior to surgery.

The primary measure of efficacy will be the gain in red cell mass in each group prior to surgery. The proportion of patients in each treatment group requiring transfusion as well as other pre-operative, peri-operative and post-operative risks will be compared. Thirty days after discharge, a survey will be administered to gauge individual patient and family acceptance of the treatments.

Expected Results Among patients scheduled for scoliosis surgery, rHuEpo treatment can significantly lower the rate of transfusion. RHuEpo treatment may lead to improved outcomes, such as decreased length of hospitalization. However, the true significance in this project lies in the investigation of rHuEpo treatment as an alternative to the PAD program that is safer and more accessible to patients and their families.

ELIGIBILITY:
Inclusion Criteria:

Scoliosis repair

Exclusion Criteria:

-

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Red cell mass at start of surgery | 21 days

SECONDARY OUTCOMES:
Requirement for blood transfusion | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Reimer, MD, Principal Investigator — The University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada